CLINICAL TRIAL: NCT01930136
Title: Long-term Effects of Caloric Restriction on Metabolic, Renal End Retinal Health in Subjectsaffected by Obesityand Type 2 Diabetes
Brief Title: Effects of Caloric Restriction in Obesity and Type 2 Diabetes
Acronym: CRESO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Istituto Superiore di Sanità (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRESO 2
Record Dates: First submitted 2013-08-23; First posted 2013-08-28 (Estimated); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: Calorie restriction; Type 2 diabetes; Obesity; Diabetic nephropathy prevention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Calorie restriction (25%) (Experimental): CR will correspond to a reduction of 25% from the total daily calorie expenditure calculated as Total Daily Energy Expenditure (TDEE) (kcal/d) using the formula from the validated Seven-Day Physical Activity Recall (PAR) Questionnaire (RMR x activity levels).
  Interventions: Behavioral: Calorie restriction (25%)
- Ad libitum health diet (Active Comparator)
  Interventions: Behavioral: Ad libitum health diet

INTERVENTIONS:
Behavioral: Calorie restriction (25%)
  Arms: Calorie restriction (25%)
Behavioral: Ad libitum health diet
  Arms: Ad libitum health diet

SUMMARY:
The study investigates whether a long-term 25% caloric restriction can prevent onset and/or progression of renal function deterioration, retinal involvement and cardiovascular complications in overweight/obese type 2 diabetic patients, trough the amelioration of concomitant metabolic abnormalities such as visceral obesity, insulin resistance, dyslipidemia, hypertension and inflammation.

The main aim of the study is therefore to evaluate the role of calorie restriction (CR) on subjects at risk of nephropathy. Secondary aims are to better understand the relationship between CR and the following aspects: renal disease and its associated metabolic abnormalities, retinopathy and cardiovascular complications, quality of life and treatment cost.

ELIGIBILITY:
Inclusion Criteria

* Age >40 years;
* Type 2 diabetes (ADA criteria);
* UAE <300 mg/24h;
* Body mass index (BMI)>27kg/m2;
* Serum creatinine < 1.2 mg/dL;
* No major changes in calorie, protein and sodium intake in the last 6 mos;
* No major changes in concomitant treatments with blood pressure, glucose or lipid lowering agents since 6 and 3 months respectively;
* Patients legally able to give written informed consent to the trial (signed and dated by the patient);
* Written informed consent.

Exclusion Criteria

* Concomitant non-diabetic renal disease or ischemic kidney disease;
* Primary or immune-mediated renal disease;
* Urinary tract obstruction or infection;
* Treatment with steroids and/or non-steroid anti-inflammatory agents;
* Treatment with thiazide or loop diuretics that, on the basis of the Investigator's judgment, might sustain hypovolemia and/or sodium depletion (with secondary kidney hypoperfusion/hypofiltration);
* Hearth failure and/or hemodynamically significant left ventricular systolic dysfunction, cirrhosis, uncontrolled hyperglycemia resulting in glycosuria, hyper/hyponatremia of any cause;
* Previous surgical procedures for weight loss;
* Previous episodes of depression, or suicide attempts;
* Chronic abuse of alcohol and drugs;
* Pregnancy, ineffective contraception or peri-menopausal age;
* Cancer or any chronic disease that might affect the completion of the study;
* Chronic obstructive pulmonary disease (COPD) in treatment with positive airway pressure;
* Unwillingness or inability to adhere to CR intervention over the entire 24-months intervention period;
* Legal incapacity and/or other circumstances rendering the patient unable to understand the nature, scope and possible consequence of the trial;
* Evidence of an uncooperative attitude;
* Any evidence that patient will not be able to complete the trial follow-up;
* Inability to fully understand the potential risks and benefits of the study.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-05-05 (Actual)

PRIMARY OUTCOMES:
The percent change in glomerular filtration rate (GFR) at month 6 versus baseline and the rate of GFR decline from month 6 to study end | At baseline, 6, 12 and 24 month

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Center for Rare Diseases, Ranica, Bergamo, Italy

REFERENCES:
- [Derived] Ruggenenti P, Cortinovis M, Trillini M, Parvanova A, Abbate M, Satriano C, Salvetti F, Bossi AC, Trevisan R, Perna A, Peracchi T, Rubis N, Diadei O, Martinetti D, Gaspari F, Fontana L, Remuzzi G; CRESO 2 Study; Organization. Long-term kidney and systemic effects of calorie restriction in overweight or obese type 2 diabetic patients (C.Re.S.O. 2 randomized controlled trial). Diabetes Res Clin Pract. 2022 Mar;185:109804. doi: 10.1016/j.diabres.2022.109804. Epub 2022 Feb 24. PMID 35219762